CLINICAL TRIAL: NCT05255575
Title: A Single Center, Prospective Clinical Trial of Intravenous Ertapenem in the Treatment of Hurley Stage II or III Hidradenitis Suppurativa
Status: Withdrawn | Type: Observational
Why Stopped: unavailable staff to support project
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Principal Investigator, Henry Ford Health System
Other Study IDs: IRB11628
Record Dates: First submitted 2022-02-16; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Ertapenem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ertapenem treatment
  Interventions: Drug: Ertapenem

INTERVENTIONS:
Drug: Ertapenem — Patients will receive ertapenem therapy.

SUMMARY:
: Treatment of chronic, recalcitrant HS presents significant challenges and frustration to both the patient and the provider. In chronic, recalcitrant HS, wide surgical excision is considered the treatment of choice.13 In 2016, Join-Lambert et al investigated the use of intravenous (IV) ertapenem in 30 patients with severe, refractory HS.14 One gram of ertapenem daily for 6 weeks followed by consolidation antibiotics for 6 months demonstrated promising results in severe, recalcitrant HS.14 These patients reported significant improvements in pain, purulent drainage, and a decrease in handicap score.14 Additionally, this technique is less invasive than surgical excision.

DETAILED DESCRIPTION:
Hidradenitis suppurativa (HS) is a chronic, socially and cosmetically debilitating disease characterized by recurrent abscesses, draining sinus tracts, and scarring with a predilection for intertriginous skin folds.1 The lesions are painful and can drain malodorous fluid, leaving patients uncomfortable and self-conscious.1 It is not surprising that HS has a high degree of morbidity or that these patients have among the lowest quality of life scores of all skin disease.2-5

The pathophysiology of HS is not fully understood. It is thought to be multifactorial.1 The primary insult is believed to be follicular occlusion with hyperkeratinization and rupture of the follicle followed by bacterial colonization and biofilm formation.1 Most cultures of HS lesions are polymicrobial and commonly grow gram positive bacteria and anaerobes.6,7 A recent study observed evidence of biofilms in chronic HS lesions.8 Lesions with bacterial biofilms respond to antibiotics initially then demonstrate resistance as the bacteria develop metabolic adaptations and produce a protective layer, the extracellular matrix.1,8 This results in persistent, recalcitrant lesions.6 Lesions are difficult to treat and present significant frustration to both the patient and the provider.

The efficacy of antibiotics in HS has been explored. Antibiotics are commonly first line therapy in HS.1,9 Rifampicin, clindamycin, and tetracycline have successfully treated HS lesions.10,11 Other effective antibiotics include: carbapenems, fluoroquinolones, and penicillins with β-lactamase inhibitors.9 Triple therapy with oral rifampin, moxifloxacin, and metronidazole has been proposed.12 Although frequently successful in early stage disease, this regimen is less effective in Hurley stage II and III HS.12 Patients with Hurley stage II and III HS rarely experience remission on antibiotics alone. In chronic, recalcitrant HS, wide surgical excision is considered the treatment of choice.13 The Hurley Staging system is commonly utilized to classify the severity of a patient's hidradenitis suppurativa. Stage 1 disease consists of one or more abscesses with no sinus tract formation or scarring. Stage 2 disease involves one or more widely separated recurrent abscesses, with formation of a sinus tract and/or scarring. Stage 3 involves multiple interconnected sinus tracts and/or abscesses throughout an anatomical area.

In 2016, Join-Lambert et al investigated the use of intravenous (IV) ertapenem in 30 patients with severe, refractory HS.14 One gram of ertapenem daily for 6 weeks followed by consolidation antibiotics for 6 months demonstrated promising results in severe, recalcitrant HS.14 These patients reported significant improvements in pain, purulent drainage, and a decrease in handicap score.14 In this study, we propose the use of ertapenem for management of Hurley stage 2 and 3 hidradenitis suppurativa as a less invasive means of treating HS. The primary endpoint will be to determine the role of ertapenem in achieving Hidradenitis Suppurativa clinical response (HiSCR) at 6 weeks. HiSCR is defined as HS Clinical Response with ≥ 50% reduction from baseline in AN (total abscess and inflammatory nodule) count with no increase in abscess or in draining fistula counts. Secondary endpoints include a change in DLQI score from baseline to the end of week, work productivity and activity impairment (WPAI) outcome from baseline to the end of week six, C- reactive protein and hemoglobin from baseline to the end of 6 weeks, the change in HS-LASI from baseline to the end of week 6, and ultrasound changes from baseline to the end of week 6.

Study Synopsis

1. PURPOSE: To determine the clinical efficacy of ertapenem for the treatment of Hurley stage 2 and 3 hidradenitis suppurativa (HS). We will be assessing safety and tolerability of this medication. We will be evaluating the effect this medication has on patient's quality of life.

2. SPECIFIC AIMS:

1. To determine the role of ertapenem in achieving Hidradenitis Suppurativa clinical response (HiSCR) at 6 weeks. HiSCR is defined as HS clinical response of ≥ 50% reduction from baseline in AN (total abscess and inflammatory nodule) count with no increase in abscess or in draining fistula counts.
2. To determine the change in DLQI score from baseline to the end of week 6.
3. To determine work impairment using the questionnaire work productivity and activity impairment- specific health problem (WPAI-SHP)
4. To determine the mean change in C- reactive protein and hemoglobin from baseline to the end of week 6.
5. To determine the change in modified HS-LASI from baseline to the end of week 6.
6. To determine ultrasound changes from baseline to the end of week 6.

3. RATIONALE FOR THE PROJECT: Treatment of chronic, recalcitrant HS presents significant challenges and frustration to both the patient and the provider. In chronic, recalcitrant HS, wide surgical excision is considered the treatment of choice.13 In 2016, Join-Lambert et al investigated the use of intravenous (IV) ertapenem in 30 patients with severe, refractory HS.14 One gram of ertapenem daily for 6 weeks followed by consolidation antibiotics for 6 months demonstrated promising results in severe, recalcitrant HS.14 These patients reported significant improvements in pain, purulent drainage, and a decrease in handicap score.14 Additionally, this technique is less invasive than surgical excision.

4. SIGNIFICANCE: This study will provide insight into the utility of ertapenem which can serve as a therapeutic, less invasive option to treat patients with refractory, Hurley stage 2 and 3 hidradenitis suppurativa.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Diagnosis of Hurley Stage II or III HS
3. Be otherwise healthy with no history of renal impairment
4. Participant must be able to understand the requirements of the study and risks involved
5. Participant must be able to sign a consent form
6. Baseline abscess and inflammatory nodule count (AN count) of 3 or more and draining fistula count of 20 or fewer
7. Unresponsive or intolerant to oral antibiotics for HS treatment as determined by the caregiver
8. Patient must be unstable with worsening inflammatory manifestations of HS
9. Diagnosis of HS for at least 6 mo (180 day) before baseline that involves at least 2 distinct anatomical areas (ex: left and right axillae)

Exclusion Criteria:

1. Any reason the investigator feels the patient should not participate in the study.
2. If a patient misses ≥ 2 consecutive study visits, the patient will be excluded from further participation in this trial.
3. History of an allergy to an antibiotic in the penicillin class.
4. If the investigator feels that a different therapeutic option would be more beneficial to the patient
5. Any other skin disease or condition (e.g. infectious or non-infectious) that may interfere with assessment of HS.
6. History of any medical condition, in the opinion of the investigator, that would put the subject at risk by participating in this study.
7. Subjects who have received biologic medications must wait 3 weeks or 21 days prior to enrollment in this research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HS patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-07-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
HiSCR | 6 weeks
  1. To determine the role of ertapenem in achieving Hidradenitis Suppurativa clinical response (HiSCR) at 6 weeks. HiSCR is defined as HS clinical response of ≥ 50% reduction from baseline in AN (total abscess and inflammatory nodule) count with no increase in abscess or in draining fistula counts.

SECONDARY OUTCOMES:
DLQI | 6 weeks
  To determine the change in DLQI score from baseline to the end of week 6
WPAI-SHP | 6 weeks
  To determine work impairment using the questionnaire work productivity and activity impairment- specific health problem (WPAI-SHP)
Labs | 6 weeks
  To determine the mean change in C- reactive protein and hemoglobin from baseline to the end of week 6.
HS-LASI | 6 weeks
  To determine the change in modified HS-LASI from baseline to the end of week 6.
Ultrasound | 6 weeks
  To determine ultrasound changes from baseline to the end of week 6.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Henry Ford Medical Center, 3031 West Grand Boulevard,, Detroit, Michigan, United States